CLINICAL TRIAL: NCT05530499
Title: Effects of Almonds on Immune Health and Responsiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Principal Investigator, Jaapna Dhillon, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2090290
Record Dates: First submitted 2022-08-30; First posted 2022-09-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diet Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Almond (Experimental): Participants in this group will be instructed to consume 57 grams of whole almonds every day for six weeks.
  Interventions: Other: Almond supplementation
- Cookie (Active Comparator): Participants in this group will be instructed to consume cookies equivalent to the energy content of 57 grams of whole almonds every day for six weeks.
  Interventions: Other: Cookie supplementation

INTERVENTIONS:
Other: Almond supplementation — Daily consumption of 57g of whole almonds
  Arms: Almond
Other: Cookie supplementation — Daily consumption of cookie snack calorically equivalent to 57 grams of whole almonds.
  Arms: Cookie

SUMMARY:
This study has the primary objective of investigating the benefits of consuming whole almonds on immune health and immune response in adults with obesity.

DETAILED DESCRIPTION:
The study is a six week, randomized, controlled, and parallel arm clinical trial in which participants will be randomized to consume either 57 grams of whole almonds daily or to consume an isocaloric cookie snack daily. Outcomes assessed will include blood and adipose immune markers, cardiometabolic biomarkers, and gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 30-45 kg/m^2
* Willingness to consume study foods
* Willing to comply with study protocol
* Consistent diet and activity patterns for 4 weeks
* Weight stable (no greater than 5 kg change over the last 3 months)
* Non-smoker > 1 year or more

Exclusion Criteria:

* Regular consumer of nuts
* Planning on getting viral vaccines during study
* Allergies to study foods (almonds, cookies)
* Illicit drug use
* Recent start of medications that affect metabolism or appetite
* Current use of medication that interfere with immune measures
* Diabetes
* Drug therapy for coronary artery disease, peripheral artery disease, congestive heart failure, or dyslipidemia
* Pregnant of lactating individuals
* Lidocaine allergies

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Change in immune and inflammatory markers | Over 6 weeks
  Lymphocytes, granulocytes, monocytes, interleukins, cytokines, etc.
Change in immune cell profile | Over 6 weeks
  Immunophenotyping

SECONDARY OUTCOMES:
Body mass | Baseline, week 3, and week 6
  Measured in kg
Body composition | Baseline, week 3, and week 6
  Fat mass and fat-free mass
Anthropometrics | Baseline, week 3, and week 6
  Waist circumference, hip circumference, thigh circumference
Glucoregulation | Baseline and week 6
  Fasting glucose concentrations
Insulinemic biomarker concentrations | Baseline and week 6
  Fasting insulin and C-peptide concentrations
Lipid profile | Baseline and week 6
  LDL, HDL, triglycerides, total cholesterol
Blood pressure | Baseline, week 3, week 6
  Diastolic and systolic blood pressure
Dietary intake | Baseline, week 1, week 2, week 3, week 4, week 5, week 6
  24 hours dietary recall and food frequency questionnaires
24 hour appetite ratings | Baseline, week 6
  24 hour appetite rating survey
Physical activity | Baseline, week 6
  Activity assessment using Actigraphs
Sleep | Baseline, week 6
  Sleep monitors and questionnaires
Transcriptomics profiles | Baseline, week 6
  RNAseq
Palatability rating of foods | Baseline, week 3, week 6
  Hedonic general labelled magnitude scale (gLMS)
Acceptance rating of foods | Baseline, week 3, week 6
  9-point food action rating scale

OTHER OUTCOMES:
Gut microbiome profile | Baseline, week 6
  16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Jaapna Dhillon, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here after deidentification (ie; text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be deposited in online repositories